CLINICAL TRIAL: NCT00227903
Title: Psychosocial Research to Improve Drug Treatment in Pregnancy (PRIDE-P)
Brief Title: Therapeutic Substance Abuse Treatment in Pregnancy - 1
Acronym: PRIDE-P
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0402026466; R01DA019135 (NIH)
Record Dates: First submitted 2005-09-27; First posted 2005-09-28 (Estimated); Results first posted 2013-08-21 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Alcohol Abuse; Cocaine Abuse; Marijuana Abuse
MeSH Terms: conditions — Alcoholism; Cocaine-Related Disorders; Marijuana Abuse | interventions — Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MI-CBT (Experimental): Motivationally-enhanced cognitive behavioral skills counseling
  Interventions: Behavioral: MI-CBT
- Brief Advice (Active Comparator): Advice and education
  Interventions: Behavioral: Brief Advice

INTERVENTIONS:
Behavioral: MI-CBT — Motivationally-enhanced cognitive behavioral skills counseling
  Arms: MI-CBT
Behavioral: Brief Advice — Advice and education
  Arms: Brief Advice

SUMMARY:
The purpose of this study is... To assess whether a behavioral treatment that combines motivational enhancement and cognitive skills training therapy (MET-CBT) is more effective than brief advice in: 1) decreasing use of a full range of psychoactive substances (e.g. marijuana, cocaine, methamphetamines, alcohol, nicotine, opioids) in pregnant substance using and dependent women; 2) decreasing HIV risk behavior; 3) improving birth outcomes (longer gestations and greater birth weight).

DETAILED DESCRIPTION:
We propose an integrated system of counseling services onsite in primary care obstetrical clinics, comparing a manualized brief advice (closely approximating "treatment as usual") to manualized motivationally enhanced cognitive behavioral therapy. Treatment providers are obstetrical nurses. Therapy patients are taught skill sets designed to enhance motivation to abstain from drugs of abuse, as well as designed to prevent relapse during the perinatal period. It is our hypothesis that therapy patients will be more successful at achieving stated study aims than those receiving brief advice.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women, age 16 or older, alcohol or illicit drug use in the past 30 days -

Exclusion Criteria:

Nonfluent in English or Spanish, pending incarceration, psychotic, cognitively unable to give informed consent, actively suicidal or homicidal, already engaged in addictions treatment, primarily addicted to nicotine or heroin.

-

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 168 (Actual)
Dates: Start 2004-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Yonkers, M.D., Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Yale-New Haven Hospital, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No
only aggregate de-identified data

REFERENCES:
- [Background] Yonkers KA, Howell HB, Allen AE, Ball SA, Pantalon MV, Rounsaville BJ. A treatment for substance abusing pregnant women. Arch Womens Ment Health. 2009 Aug;12(4):221-7. doi: 10.1007/s00737-009-0069-2. Epub 2009 Apr 7. PMID 19350369
- [Background] Hine CE, Howell HB, Yonkers KA. Integration of medical and psychological treatment within the primary health care setting. Soc Work Health Care. 2008;47(2):122-34. doi: 10.1080/00981380801970244. PMID 18956504
- [Background] Yonkers KA, Gotman N, Kershaw T, Forray A, Howell HB, Rounsaville BJ. Screening for prenatal substance use: development of the Substance Use Risk Profile-Pregnancy scale. Obstet Gynecol. 2010 Oct;116(4):827-833. doi: 10.1097/AOG.0b013e3181ed8290. PMID 20859145
- [Background] Quesada O, Gotman N, Howell HB, Funai EF, Rounsaville BJ, Yonkers KA. Prenatal hazardous substance use and adverse birth outcomes. J Matern Fetal Neonatal Med. 2012 Aug;25(8):1222-7. doi: 10.3109/14767058.2011.602143. Epub 2012 May 11. PMID 22489543
- [Result] Yonkers KA, Forray A, Howell HB, Gotman N, Kershaw T, Rounsaville BJ, Carroll KM. Motivational enhancement therapy coupled with cognitive behavioral therapy versus brief advice: a randomized trial for treatment of hazardous substance use in pregnancy and after delivery. Gen Hosp Psychiatry. 2012 Sep-Oct;34(5):439-49. doi: 10.1016/j.genhosppsych.2012.06.002. Epub 2012 Jul 12. PMID 22795046
- [Derived] Xu X, Yonkers KA, Ruger JP. Economic evaluation of a behavioral intervention versus brief advice for substance use treatment in pregnant women: results from a randomized controlled trial. BMC Pregnancy Childbirth. 2017 Mar 7;17(1):83. doi: 10.1186/s12884-017-1260-5. PMID 28270105
- [Derived] Forray A, Gotman N, Kershaw T, Yonkers KA. Perinatal smoking and depression in women with concurrent substance use. Addict Behav. 2014 Apr;39(4):749-56. doi: 10.1016/j.addbeh.2013.12.008. Epub 2013 Dec 17. PMID 24447885

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between June 2006 and September 2009, with follow-up concluding in July 2010. Women were screened and recruited while attending obstetrical appointments in two hospital-based reproductive health clinics in New Haven and Bridgeport, CT.
Pre-assignment Details: 13 women who were consented to the trial and provisionally were found to be eligible either declined or failed to complete intake, 1 had an incomplete intake and 1 was found to be ineligible at intake
Period: Overall Study
Arm/Group | Brief Advice | MI-CBT
Started | 91 | 92
Received ≥ 1 Follow-up Assessment | 86 (1 participant did not receive any treatment sessions.) | 82 (4 participants did not receive any treatment sessions.)
Completed | 86 (Participants with at least 1 follow-up assessment were analyzed) | 82 (Participants with at least 1 follow-up assessment were analyzed)
Not Completed | 5 | 10
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Subject moved out of area | 1 | 2
Not completed — Lost to Follow-up | 1 | 3
Not completed — Miscarriage | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis excluded women with no follow-up assessments.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brief Advice | MI-CBT | Total
Number analyzed (Participants) | 86 | 82 | 168
Age, Customized [Number; unit: participants]
  <20 years | 13 | 16 | 29
  20-34 years | 65 | 61 | 126
  >35 years | 8 | 5 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 82 | 168
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — Participants could indicate more than one race/ethnicity category. All results were counted and categorized, leading to a total count greater than the number baseline participants.
  participants
    White | 17 | 19 | 36
    Black | 47 | 42 | 89
    Hispanic | 24 | 19 | 43
    Other | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 86 | 82 | 168
Education (years) [Number; unit: participants]
  <12 | 26 | 32 | 58
  12 | 31 | 35 | 66
  13-15 | 23 | 14 | 37
  16+ | 6 | 1 | 7
Parity [Count of Participants; unit: Participants] — Parity defined as number of previous births
  Participants
    0 | 35 | 31 | 66
    1 | 27 | 25 | 52
    2+ | 24 | 26 | 50
Gestational age at intake [Number; unit: participants]
  Weeks 1-8 | 5 | 3 | 8
  Weeks 9-16 | 25 | 28 | 53
  Weeks 17-24 | 31 | 27 | 58
  Weeks 25 or later | 25 | 24 | 49
Prenatal care initiation [Number; unit: participants]
  Weeks 1-8 | 21 | 23 | 44
  Weeks 9-16 | 47 | 40 | 87
  Weeks 17-24 | 13 | 10 | 23
  Week 25 or later | 4 | 5 | 9
  Unknown | 1 | 4 | 5
Site [Number; unit: participants]
  Bridgeport Hospital | 22 | 25 | 47
  Yale New Haven Hospital | 64 | 57 | 121
MINI drug or alcohol abuse or dependence [Number; unit: participants]
  Participants diagnosed with abuse or dependence | 28 | 19 | 47
  Participants without such a diagnosis | 58 | 63 | 121
Past-month use [Number; unit: participants] — Participants could indicate use of more than one substance in the past month. All results were counted and categorized, leading to a total count greater than the number of baseline participants.
  participants
    Alcohol (any) | 33 | 19 | 52
    Alcohol (intoxication) | 7 | 9 | 16
    Heroin | 1 | 3 | 4
    Methadone | 5 | 8 | 13
    Opiates (excluding methadone) | 6 | 4 | 10
    Barbiturates | 0 | 0 | 0
    Sedatives | 5 | 1 | 6
    Cocaine | 11 | 7 | 18
    Amphetamines | 1 | 0 | 1
    Marijuana | 40 | 34 | 74
    Hallucinogens | 2 | 1 | 3
    Inhalants | 0 | 0 | 0
Primary Drug [Number; unit: participants] — Primary drug was determined by combining a) self-reported recent use of substances and b) preferred substance according to the subject. If the participant used only one substance in the past 28 days, it was designated as primary. If the woman used more than one or did not endorse use of a substance in the prior 28 days, we used patient-identified primary drug. Subjects who reported more than one drug as primary were classified as "other" regardless of substances endorsed.
  participants
    Alcohol | 25 | 26 | 51
    Cocaine | 15 | 14 | 29
    Marijuana | 40 | 37 | 77
    Other | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Days Used Drugs or Alcohol
Time Frame: intake to delivery, an average of 21 weeks
Population: all randomized participants
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 86 | 82
percentage of days
  Intake | 18 (27) | 21 (34)
  Delivery | 6 (17) | 7 (22)
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; We estimated that 110 people with 10% attrition would provide 80% power; Test type: Superiority or Other; p = 0.88, Mixed Models Analysis — Not corrected for multiple comparison; 2 degrees of freedom

2. Secondary Outcome: Incidence of Preterm Births
Time Frame: At delivery
Population: A singleton live birth occurred in 163 subjects, and 5 had twins. Data was collected from the 84 women of the Brief Advice category and the 79 women of the MI-CBT category who had singleton live births.
Measure: Number; unit: preterm births
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 84 | 79
preterm births | 17 | 8
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.08, Fisher Exact

3. Primary Outcome: Percentage of Days Used Drugs or Alcohol
Time Frame: delivery to 3 months post-delivery
Population: all randomized participants with data from delivery and 3 months post-delivery
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 83 | 80
percentage of days
  Delivery | 6 (17) | 7 (22)
  3 months post-delivery | 14 (25) | 13 (24)
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; We estimated that 110 people with 10% attrition would provide 80% power; Test type: Superiority or Other; p = 0.88, Mixed Models Analysis — Not corrected for multiple comparison; 2 degrees of freedom

4. Secondary Outcome: Incidence of Low Birth Weight
Time Frame: At delivery
Population: Only singleton live births, which occurred in 163 subjects, were analyzed. Three of the women in the MI-CBT group had an infant of unknown birth weight, and were not included in analysis.
Measure: Number; unit: low weight births
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 84 | 76
low weight births | 17 | 11
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.41, Fisher Exact

5. Secondary Outcome: Proportion of Participants Abstinent From Both Drugs and Alcohol (28 Days Prior to Assessment) According to Self-report
Time Frame: intake to delivery, an average of 21 weeks
Population: All randomized participants
Measure: Number; unit: proportion of participants
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 86 | 82
proportion of participants
  Intake | 0.41 | 0.49
  Delivery | 0.75 | 0.76
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.79, Regression, Logistic; Odds Ratio (OR) = .77, 95% CI 2-sided [0.36 to 1.67]

6. Secondary Outcome: Proportion of Participants Abstinent From Both Drugs and Alcohol (28 Days Prior to Assessment) According to Self-report
Time Frame: Delivery to 3 months post-delivery
Population: All randomized participants with data available from the time frame.
Measure: Number; unit: proportion of participants
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 83 | 80
proportion of participants
  Delivery | 0.75 | 0.76
  3 months post-delivery | 0.38 | 0.41
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.79, Regression, Logistic; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.42 to 2.62]

7. Secondary Outcome: Proportion of Participants Abstinent From Drugs (i.e., Marijuana, Cocaine or Opioids) According to Urine
Time Frame: intake to delivery, an average of 21 weeks
Population: All randomized participants for whom urine test data was available.
Measure: Number; unit: proportion of participants
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 80 | 81
proportion of participants
  Intake | 0.54 | 0.56
  Delivery | 0.84 | 0.84
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.88, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.34 to 2.72]

8. Secondary Outcome: Proportion of Participants Abstinent From Drugs According to Urine
Description: Based on urine tests for marijuana, cocaine, or opioids
Time Frame: Delivery to 3 months post-delivery
Population: All randomized participants for whom urine data was available during the time frame.
Measure: Number; unit: proportion of participants
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 51 | 55
proportion of participants
  Delivery | 0.84 | 0.84
  3 months post-delivery | 0.52 | 0.59
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.88, Regression, Logistic; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.57 to 2.57]

9. Secondary Outcome: Proportion of Participants Abstinent From Both Drugs and Alcohol According to Combined Self-report and Urine
Description: Based on urine tests for marijuana, cocaine or opioids.
Time Frame: intake to delivery, an average of 21 weeks
Population: All randomized participants with both self-report and urine data available.
Measure: Number; unit: proportion of participants
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 80 | 81
proportion of participants
  Intake | 0.33 | 0.43
  Delivery | 0.76 | 0.75
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.50, Regression, Logistic; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.32 to 1.84]

10. Primary Outcome: Percentage of Days That Participants (Without a Baseline Diagnosis of Drug Abuse or Dependence) Used Drugs or Alcohol
Time Frame: intake to delivery, an average of 21 weeks
Population: All randomized participants without a baseline diagnosis of drug use or dependence.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 58 | 63
percentage of days
  Intake | 14 (25) | 15 (27)
  Delivery | 4 (11) | 6 (20)
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.10, Mixed Models Analysis

11. Primary Outcome: Percentage of Days That Participants (Without a Baseline Diagnosis of Drug Abuse or Dependence) Used Drugs or Alcohol
Time Frame: Delivery to 3 months post-delivery
Population: All randomized participants without a baseline diagnosis for drug abuse or dependence with data available for time frame.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 55 | 62
percentage of days
  Delivery | 4 (11) | 6 (20)
  3 months post-delivery | 11 (20) | 14 (27)
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.10, Mixed Models Analysis

12. Primary Outcome: Percentage of Days That Participants (With a Baseline Diagnosis of Drug Abuse or Dependence) Used Drugs or Alcohol
Time Frame: intake to delivery, an average of 21 weeks
Population: All randomized participants with a baseline diagnosis for drug abuse or dependence.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 28 | 19
percentage of days
  Intake | 27 (29) | 40 (45)
  Delivery | 10 (25) | 13 (28)
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.10, Mixed Models Analysis

13. Primary Outcome: Percentage of Days That Participants (With a Baseline Diagnosis of Drug Abuse or Dependence) Used Drugs or Alcohol
Time Frame: Delivery to 3 months post-delivery
Population: All randomized participants with a baseline diagnosis of drug abuse or dependence and data available for the time frame.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 28 | 18
percentage of days
  Delivery | 10 (25) | 13 (28)
  3 months post-delivery | 18 (32) | 8 (8)
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.10, Mixed Models Analysis

14. Secondary Outcome: Proportion of Participants Abstinent From Both Drugs and Alcohol According to Combined Self-report and Urine
Description: Based on urine tests for marijuana, cocaine, or opioids.
Time Frame: Delivery to 3 months post-delivery
Population: All randomized participants with both self-report and urine data available during the time frame.
Measure: Number; unit: proportion of participants
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 51 | 55
proportion of participants
  Delivery | 0.76 | 0.75
  3 months post-delivery | 0.34 | 0.33
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.50, Regression, Logistic; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.27 to 2.11]

15. Secondary Outcome: Proportion of Participants (Without a Baseline Diagnosis of Drug Abuse or Dependence) Abstinent From Both Drugs and Alcohol (28 Days Prior to Assessment) According to Self-report
Time Frame: intake to delivery, an average of 21 weeks
Population: All randomized participants without a baseline diagnosis of drug abuse or dependence.
Measure: Number; unit: proportion of participants
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 58 | 63
proportion of participants
  Intake | 0.50 | 0.52
  Delivery | 0.76 | 0.81
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.07, Regression, Logistic; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.44 to 3.14]

16. Secondary Outcome: Proportion of Participants (Without a Baseline Diagnosis of Drug Abuse or Dependence) Abstinent From Both Drugs and Alcohol (28 Days Prior to Assessment) According to Self-report
Time Frame: Delivery to 3 months post-delivery
Population: All randomized participants without a baseline diagnosis of drug abuse or dependence with data available for the time frame.
Measure: Number; unit: proportion of participants
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 55 | 62
proportion of participants
  Delivery | 0.76 | 0.81
  3 months post-delivery | 0.28 | 0.44
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.07, Regression, Logistic; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.47 to 4.52]

17. Secondary Outcome: Proportion of Participants (With a Baseline Diagnosis of Drug Abuse or Dependence) Abstinent From Both Drugs and Alcohol (28 Days Prior to Assessment) According to Self-report
Time Frame: intake to delivery, an average of 21 weeks
Population: All randomized participants with a baseline diagnosis of drug abuse or dependence.
Measure: Number; unit: proportion of participants
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 28 | 19
proportion of participants
  Intake | 0.21 | 0.37
  Delivery | 0.71 | 0.61
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.07, Regression, Logistic; Odds Ratio (OR) = 0.28, 95% CI 2-sided [0.08 to 1.02]

18. Secondary Outcome: Proportion of Participants (With a Baseline Diagnosis of Drug Abuse or Dependence) Abstinent From Both Drugs and Alcohol (28 Days Prior to Assessment) According to Self-report
Time Frame: Delivery to 3 months post-delivery
Population: All randomized participants with a baseline diagnosis of drug abuse or dependence and data available for the time frame.
Measure: Number; unit: proportion of participants
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 28 | 18
proportion of participants
  Delivery | 0.71 | 0.61
  3 months post-delivery | 0.54 | 0.31
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.07, Regression, Logistic; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.10 to 3.90]

19. Secondary Outcome: Proportion of Participants (Without a Baseline Diagnosis of Drug Abuse or Dependence) Abstinent From Drugs According to Urine
Description: Based on urine tests for marijuana, cocaine or opioids.
Time Frame: intake to delivery, an average of 21 weeks
Population: All randomized participants without a baseline diagnosis for drug abuse or dependence and with urine data.
Measure: Number; unit: proportion of participants
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 52 | 62
proportion of participants
  Intake | 0.56 | 0.60
  Delivery | 0.82 | 0.85
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.91, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.32 to 4.20]

20. Secondary Outcome: Proportion of Participants (Without a Baseline Diagnosis of Drug Abuse or Dependence) Abstinent From Drugs According to Urine
Description: Based on urine tests for marijuana, cocaine or opioids.
Time Frame: Delivery to 3 months post-delivery
Population: All randomized participants without a baseline diagnosis of drug abuse or dependence and urine data during the time frame.
Measure: Number; unit: proportion of participants
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 33 | 46
proportion of participants
  Delivery | 0.82 | 0.85
  3 months post-delivery | 0.46 | 0.58
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.91, Regression, Logistic; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.35 to 5.07]

21. Secondary Outcome: Proportion of Participants (With a Baseline Diagnosis of Drug Abuse or Dependence) Abstinent From Drugs According to Urine
Description: Based on urine tests for marijuana, cocaine or opioids.
Time Frame: intake to delivery, an average of 21 weeks
Population: All randomized participants with a baseline diagnosis of drug abuse or dependence and urine data.
Measure: Number; unit: proportion of participants
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 28 | 19
proportion of participants
  Intake | 0.50 | 0.42
  Delivery | 0.89 | 0.78
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.91, Regression, Logistic; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.14 to 5.23]

22. Secondary Outcome: Proportion of Participants (With a Baseline Diagnosis of Drug Abuse or Dependence) Abstinent From Drugs According to Urine
Description: Based on urine tests for marijuana, cocaine or opioids.
Time Frame: Delivery to 3 months post-delivery
Population: All randomized participants with a baseline diagnosis of drug abuse or dependence and urine data.
Measure: Number; unit: proportion of participants
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 18 | 9
proportion of participants
  Delivery | 0.89 | 0.78
  3 months post-delivery | 0.60 | 0.63
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.91, Regression, Logistic; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.21 to 7.12]

23. Secondary Outcome: Proportion of Participants (Without a Baseline Diagnosis of Drug Abuse or Dependence) Abstinent From Both Drugs and Alcohol According to Combined Self-report and Urine
Description: Based on urine tests for marijuana, cocaine or opioids.
Time Frame: intake to delivery, an average of 21 weeks
Population: All randomized participants without a baseline diagnosis of drug abuse or dependence, and with both self-report and urine data.
Measure: Number; unit: proportion of participants
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 52 | 62
proportion of participants
  Intake | 0.42 | 0.47
  Delivery | 0.76 | 0.76
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = .04, Regression, Logistic; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.46 to 3.55]

24. Secondary Outcome: Proportion of Participants (Without a Baseline Diagnosis of Drug Abuse or Dependence) Abstinent From Both Drugs and Alcohol According to Combined Self-report and Urine
Description: Based on urine tests for marijuana, cocaine or opioids
Time Frame: Delivery to 3 months post-delivery
Population: All randomized participants without a baseline diagnosis of drug abuse or dependence, and with both self-report and urine data for the time frame.
Measure: Number; unit: proportion of participants
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 33 | 46
proportion of participants
  Delivery | 0.76 | 0.76
  3 months post-delivery | 0.23 | 0.35
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.04, Regression, Logistic; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.35 to 4.17]

25. Secondary Outcome: Proportion of Participants (With a Baseline Diagnosis of Drug Abuse or Dependence) Abstinent From Both Drugs and Alcohol According to Combined Self-report and Urine
Description: Based on urine tests for marijuana, cocaine or opioids
Time Frame: intake to delivery, an average of 21 weeks
Population: All randomized participants with a baseline diagnosis for drug abuse or dependence, and with both self-report and urine data.
Measure: Number; unit: proportion of participants
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 28 | 19
proportion of participants
  Intake | 0.14 | 0.32
  Delivery | 0.78 | 0.67
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.04, Regression, Logistic; Odds Ratio (OR) = 0.25, 95% CI 2-sided [0.04 to 1.63]

26. Secondary Outcome: Proportion of Participants (With a Baseline Diagnosis of Drug Abuse or Dependence) Abstinent From Both Drugs and Alcohol According to Combined Self-report and Urine
Description: Based on urine tests for marijuana, cocaine or opioids
Time Frame: Delivery to 3 months post-delivery
Population: All randomized participants with a baseline diagnosis of drug abuse or dependence, and with both self-report and urine data for the time frame.
Measure: Number; unit: proportion of participants
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 18 | 9
proportion of participants
  Delivery | 0.78 | 0.67
  3 months post-delivery | 0.52 | 0.25
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.04, Regression, Logistic; Odds Ratio (OR) = 0.40, 95% CI 2-sided [0.04 to 3.74]

27. Other Pre Specified Outcome: Adequacy of Received Services
Description: Based on prenatal care attendance: the percent of visits attended after prenatal care initiation, accounting for time of delivery. Attendance was rated according to the Kotelchuck Adequacy of Prenatal Care Index. Only the normally scheduled prenatal car visits were included.
Time Frame: After prenatal care initiation
Population: All randomized participants, 6 women had unkown attendance.
Measure: Number; unit: participants
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 86 | 82
participants
  Inadequate (0-49% attendance) | 2 | 2
  Intermediate (50%-79% attendance) | 7 | 13
  Adequate (80%-109% attendance) | 24 | 33
  Adequate plus (110+%) | 51 | 30
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p = 0.01, Cochran-Mantel-Haenszel

28. Other Pre Specified Outcome: Attendance of Treatment Outside the Study
Description: The number of patients who attended outside treatment in the 30 days prior to each assessment.
Time Frame: 30 days prior to assessment
Population: all randomized participants with data availabe at time frames
Measure: Number; unit: participants
Arm/Group | Brief Advice | MI-CBT
Number analyzed (Participants) | 86 | 82
participants
  Participants who attended prior to delivery | 4 | 6
  Participants who attended prior to 3 months post | 9 | 6
Statistical Analysis 1: Comparison: Brief Advice vs MI-CBT; Test type: Superiority or Other; p > 0.05, Chi-squared

ADVERSE EVENTS:
Arm/Group | Brief Advice | MI-CBT
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/82
Other Adverse Events (participants affected / at risk) | 0/86 | 0/82

LIMITATIONS AND CAVEATS:
Did not acheive desired sample size; results were averaged across substances; women were not seeking substance abuse treatment (i.e. they were attending for prenatal care); treatment was brief

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No